CLINICAL TRIAL: NCT01435356
Title: A Randomized, Double Blind, Placebo Controlled Phase II Trial to Evaluate the Safety and Efficacy of recMAGE-A3 + AS15 ASCI in Patients With MAGE-A3 Positive Muscle Invasive Bladder Cancer After Cystectomy
Brief Title: Safety and Efficacy Study of MAGE-A3 + AS-15 in Patients With Muscle-invasive Bladder Cancer After Cystectomy
Acronym: MAGNOLIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: European Association of Urology Research Foundation (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EAU RF 2010-01; NTR2846 (Registry Identifier: NTR); 2010-024355-85 (EudraCT Number)
Record Dates: First submitted 2011-09-02; First posted 2011-09-16 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Urinary Bladder neoplasms; Lymphoproliferative Disorders; Immune System Diseases; Cystectomy; Adjuvants, Immunologic; Immunologic Factors
MeSH Terms: conditions — Urinary Bladder Neoplasms; Lymphoproliferative Disorders; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- recMage-A3 + AS15 ASCI (Active Comparator): MAGE-A3 positive patients treated with recMAGE-A3 + AS15 ASCI
  Interventions: Biological: recMAGE-A3 + AS15 ASCI
- Placebo (Placebo Comparator): MAGE-A3 positive patients treated with placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: recMAGE-A3 + AS15 ASCI — 5 doses were administered (intramuscular) at 3-week intervals followed by 8 doses administered at 3-month intervals for a total maximum duration of study treatment administration of 27 months
  Arms: recMage-A3 + AS15 ASCI
Biological: Placebo — 5 doses were administered (intramuscular) at 3-week intervals followed by 8 doses administered at 3-month intervals for a total maximum duration of study treatment administration of 27 months
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial was to demonstrate the benefit of the immunotherapeutic product recMAGE-A3 + AS-15 given to patients with bladder cancer after removal of the bladder. A course of 13 injections was administered over 27 months.

DETAILED DESCRIPTION:
This study assessed an investigational treatment for patients with Muscle Invasive Bladder Cancer in whom the urinary bladder had been surgically removed. The investigational treatment aimed to increase the body's immune response to a specific antigen expressed by the cancer. The tumour tissue was first tested whether it expressed the MAGE-A3 antigen.

The MAGNOLIA study was open to male and female patients with pathologically confirmed muscle invasive transitional cell carcinoma of the urinary bladder with expression of the antigen MAGE-A3 with or without limited lymph node involvement who had no evidence of disease after surgery confirmed with imaging procedures (scans CT/MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Aged greater than or equal to 18 years at the time ICF is signed, either sex.
2. Histologically confirmed (after cystectomy or if needed transurethral resection) urothelial carcinoma of the bladder which is MAGE-A3 positive.
3. Written informed consent for tissue sampling, the mandatory analyses and for the complete study has been obtained prior to the performance of any other protocol-specific procedure.
4. TNM classification at pathological examination of surgically removed specimen: Stage T2,3 N0 or N1 or N2 and M0 disease or Stage T4 N0 M0 disease.
5. The patient is free of residual disease and free of metastasis, as confirmed by a negative baseline Computer Tomogram (CT scan) or Magnetic Resonance Imaging (MRI) of the pelvis, abdomen and chest no more than 13 weeks prior to randomization. Other examinations should be performed as clinically indicated.
6. Patient is fully recovered from surgery within 13 weeks following cystectomy. For patients who receive adjuvant chemotherapy, the patient is fully recovered within 3-6 weeks following chemotherapy.
7. The patient must have adequate bone-marrow reserve, defined as an absolute neutrophil count 1.0 x 109/L, and a platelet count ≥ 75 x 109/L, adequate renal function, defined as a serum creatinine ≤ 1.5 times the Upper Limit of Normal (ULN), and adequate hepatic function, defined as a Total bilirubin ≤ 1.5 times the ULN, and a Alanine transaminase (ALAT) and Aspartate Transaminase (ASAT) ≤ 2.5 times the ULN as assessed by standard laboratory criteria.
8. World Health Organization (WHO) performance status 0 - 1 at the time of randomization.
9. If the patient is female, she must be of non-childbearing potential, i.e. have a current tubal ligation, hysterectomy, ovariectomy or be post menopausal, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to administration of study treatment, have a negative pregnancy test and continue such precautions during all study treatment period and for 2 months after completion of the injection series.
10. The patient should be affiliated to health insurance or benefit of such an insurance

Exclusion Criteria:

1. The patient has previous or concomitant malignancies at other sites except effectively treated non-melanoma skin cancer, cervical carcinoma in situ, incidental localised prostatic carcinoma or effectively treated malignancy that has been in remission for over 5 years.
2. The patient has received any anti cancer systemic treatment, including immunotherapy (local intravesical BCG is allowed), chemotherapy, except:

   * For the treatment of previous malignancies as allowed by the protocol (i.e., non-melanoma skin cancer, cervical carcinoma in situ, incidental localised prostatic carcinoma or effectively treated malignancy that has been in remission for over 5 years).
   * For the treatment with neo-adjuvant chemotherapy for their muscle invasive bladder cancer
   * For the treatment with adjuvant cisplatinum-based chemotherapy for their muscle invasive bladder cancer
3. The patient has received radiotherapy of the abdominal or pelvic region, within 6 months prior to randomization.
4. Women who are pregnant or breast feeding.
5. The patient has a known infection with human immunodeficiency virus (HIV) or chronic hepatitis B or C.
6. The patient has a history of allergic disease or reactions likely to be exacerbated by any component of the study investigational product.
7. The patient has any confirmed or suspected immunosuppressive or immunodeficient condition or potential immune-mediated diseases as. Patients with vitiligo are not excluded to participate in the trial.
8. Patient has received a major organ allograft.
9. The patient requires concomitant treatment with systemic corticosteroids, or any other immunosuppressive agents. Note: the use of prednisone, or equivalent, < 0,125 mg/kg/day (absolute maximum 10 mg/day), or inhaled corticosteroids or topical steroids is permitted.
10. The patient has received any investigational or non-registered medicinal product other than the study medication within the 30 days preceding the first dose of study medication, or plans to receive such a drug during the study.
11. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures.
12. The patient has other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk. For example, but not limited to: uncontrolled congestive heart failure or uncontrolled hypertension, unstable heart disease (coronary heart disease or myocardial infarction), uncontrolled arrhythmia or patients taking anticoagulant treatment or having a coagulation disorder.
13. The patient uses alternative treatments eg. plant extracts.
14. Adults under legal supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter FA Mulders, Prof,PhD,MD, Principal Investigator — EAU Research Foundation
Locations (50):
- Czechia (4):
  - Faculty teaching Hospital in Plzen, Pilsen
  - Hospital Motol, Prague
  - Thomayerova nemocnice, Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
- France (5):
  - Institut Bergonié, Bordeaux
  - Hôpital Huriez, Lille
  - Hôpital Edouard Herriot, Lyon
  - Institut Curie, Paris
  - Hôpital Rangueil, Toulouse
- Germany (11):
  - Universitätsklinikum Aachen, Aachen
  - Universitätsklinikum C.-G. Carus Dresden, Dresden
  - Heinrich-Heine University, Düsseldorf
  - Waldkrankenhaus St. Marien gGmbH, Erlangen
  - Universitätsklinikum Giessen, Giessen
  - Universitätsklinikum Jena, Jena
  - Universitätsmedizin, Mannheim
  - Universitätsklinikum Marburg, Marburg
  - Klinikum rechts der Isar der TU München, München
  - Universitätklinikum Rostock, Rostock
  - Universitätsklinikum Tübingen, Tübingen
- Italy (5):
  - Universitaria Policlinico Consorziale di Bari, Bari
  - Università Vita e Saluta, Milan
  - Ospedaliera di Perugia, Perugia
  - Universitaria Pisana, Pisa
  - Università di Roma, La Sapienza, Rome
- Netherlands (3):
  - NKI, Amsterdam
  - St Antoniusziekenhuis, Nieuwegein
  - RadboudUMC, Nijmegen
- Poland (3):
  - Kliniczny Dzial Urologii Swietokrzyskiego Centrum Onkologii, Kielce
  - Medical University of Warsaw, Warsaw
  - Oddzial Urologii Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw
- Romania (2):
  - Fundeni Clinical Institute, Bucharest
  - Clinical County Emergency Hospital Craiova, Craiova
- Russia (5):
  - Federal State Budget Institution "Scientific Research Institute of Urology" of the Ministry of Healthcare and Social Development of the Russian Federation, Moscow
  - Federal State Institution "Moscow Research Oncology Institute named after P.A. Gertsen" of the Ministry of Healthcare and Social Development of the Russian Federation, Moscow
  - Institution of the Russian Academy of Medical Science Russian Oncology Research Center named after N.N. Blokhin of RAMS, Moscow
  - Municipal Budget Institution of Health Care "Clinical Diagnostic Center "Zdorovie" of Rostov-on-Don city", Rostov-on-Don
  - Saint Petersburg State Institution of Health Care "City Multi-Field Hospital #2", Saint Petersburg
- Spain (11):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Principe de Asturias, Alcalá de Henares
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - Fundación Puigvert, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital 12 de Octubre, Fundación de Investigación Biomédica, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Infanta Sofia, San Sebastián de los Reyes
- Kyiv City Clinical Oncology Hospital, Kiev, Ukraine

REFERENCES:
- [Background] Colombel M, Heidenreich A, Martinez-Pineiro L, Babjuk M, Korneyev I, Surcel C, Yakovlev P, Colombo R, Radziszewski P, Witjes F, Schipper R, Mulders P, Witjes WP. Perioperative chemotherapy in muscle-invasive bladder cancer: overview and the unmet clinical need for alternative adjuvant therapy as studied in the MAGNOLIA trial. Eur Urol. 2014 Mar;65(3):509-11. doi: 10.1016/j.eururo.2013.10.056. Epub 2013 Nov 11. PMID 24268503
- See also: Pubmed — https://www.ncbi.nlm.nih.gov/pubmed/24268503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 83 patients were randomised, 52 for recMAGE-A3 +AS15 and 31 for placebo treatment. 6 patients did not start treatment due to ineligibility (4 for recMAGE-A3 +AS15 and 2 for placebo treatment).
Groups:
- recMage-A3 + AS15 ASCI: MAGE A3 positive patients treated with recMAGE-A3 + AS15 ASCI
  recMAGE-A3 + AS15 ASCI: 5 doses were administered (intramuscular) at 3-week intervals followed by 8 doses administered at 3-month intervals for a total maximum duration of study treatment administration of 27 months
Period: Overall Study
Arm/Group | recMage-A3 + AS15 ASCI | Placebo
Started | 48 | 29
Completed | 16 | 5
Not Completed | 32 | 24
Not completed — Adverse Event | 2 | 0
Not completed — Disease progression/recurrence | 17 | 10
Not completed — Protocol Violation | 0 | 1
Not completed — Study Discontinuation, amendment 4 | 5 | 11
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Facial palsy | 1 | 0
Not completed — IC withdrawal due to study cancellation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Patient decision | 3 | 0
Not completed — Patient moved to another city | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Total Treated population included all treated patients, i.e. all patients with at least one documented dose of study treatment (ASCI or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | recMage-A3 + AS15 ASCI | Placebo | Total
Number analyzed (Participants) | 48 | 29 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.4) | 65.5 (9.6) | 65.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 40 | 21 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 4 | 7 | 11
  Czechia | 6 | 1 | 7
  Poland | 1 | 0 | 1
  Italy | 0 | 2 | 2
  France | 9 | 3 | 12
  Germany | 7 | 3 | 10
  Russia | 3 | 2 | 5
  Spain | 18 | 11 | 29
T-category of bladder cancer at diagnosis [Count of Participants; unit: Participants] — Population: T2 (tumor invades muscle), T3 (tumor invades perivesical tissue), T4 (tumor invades any of the following: prostate, uterus, vagina, pelvic wall, abdominal wall).
  Participants
    T2 | 22 | 13 | 35
    T3 | 21 | 13 | 34
    T4 | 5 | 3 | 8
N-category classification of bladder cancer at diagnosis [Count of Participants; unit: Participants] — N0: No regional lymph node metastasis N1: Metastasis in a single lymph node 2 cm or less in greatest dimension N2: Metastasis in n a single lymph node more than 2 cm but not more than 5 cm in greatest dimension, or multiple lymph nodes, none more than 5 cm in greatest dimension.
  Participants
    N0 | 36 | 22 | 58
    N1 | 7 | 4 | 11
    N2 | 5 | 3 | 8
M-category of bladder cancer at diagnosis [Count of Participants; unit: Participants] — M0: No distant metastasis M1: Distant metastasis
  Participants
    M0 | 48 | 29 | 77
    M1 | 0 | 0 | 0
Dominant Histological Type [Count of Participants; unit: Participants]
  transitional (urothelial) cell carcinoma | 43 | 29 | 72
  squamous cell carcinoma | 3 | 0 | 3
  adenocarcinoma | 1 | 0 | 1
  Not available | 1 | 0 | 1
Mean weight [Mean (Standard Deviation); unit: kg] | 73.5 (13.3) | 75.1 (12.8) | 74.1 (13.4)
Mean Height [Mean (Standard Deviation); unit: cm] | 172 (7.2) | 169 (9.8) | 171 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival
Description: To evaluate of the clinical efficacy in terms of Disease Free Survival of treatment versus placebo in the overall population of patients with bladder cancer with MAGE-A3 expression after cystectomy. Disease Free Survival is the time from randomization to either the date of first recurrence of the disease or the date of death (whatever the cause), whichever occurred first. Types of recurrence considered as an event included loco-regional and distant metastases. In addition, any death occurring without prior documentation of tumor recurrence was considered as an event (and was not censored in the statistical analysis) as this approach is less prone to introduce bias.
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | recMage-A3 + AS15 ASCI | Placebo
Number analyzed (Participants) | 48 | 29
months | 27.5 [22.7 to 32.3] | 19.8 [15.7 to 23.9]

2. Secondary Outcome: Overall Survival
Description: To evaluate overall survival in the overall study population. Overall Survival was defined as the interval from randomization to the date of death, irrespective of the cause of death; patients still alive were censored at the date of the last assessment.
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | recMage-A3 + AS15 ASCI | Placebo
Number analyzed (Participants) | 48 | 29
months | 35.5 [32.1 to 38.8] | 24.1 [21 to 27.2]

3. Secondary Outcome: Disease-free Specific Survival
Description: To evaluate Disease-free specific survival in the overall population.Disease-free specific survival was defined as the interval from randomization to the date of first recurrence of disease or date of death due to bladder carcinoma, whichever occurred first. Patients without recurrence or death were censored at the date of last assessment. Patients without recurrence who died from another cause were censored at the date of death.
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | recMage-A3 + AS15 ASCI | Placebo
Number analyzed (Participants) | 48 | 29
months | 27.5 [22.7 to 32.3] | 19.8 [15.7 to 23.9]

4. Secondary Outcome: Distant Metastasis-free Survival
Description: To evaluate Distant metastasis-free survival in the overall study population. Distant metastasis-free survival was defined as the interval from randomization to the date of first distant metastasis or date of death, whichever occurred first. Patients alive and without distant metastasis were censored at the date of last assessment.
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | recMage-A3 + AS15 ASCI | Placebo
Number analyzed (Participants) | 48 | 29
months | 31.5 [27.2 to 35.9] | 21.4 [17.5 to 25.2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 5 years (between Informed Consent First Patient and Last Visit Last Patient).
Description: It was pre-specified in the Protocol that Foreseeable AEs and SAEs specifically related to the cystectomy prior to first study treatment administration will not be considered as "Adverse Events". It was left to the investigator to asses the relation between the (S)AEs and the cystectomy. Progression/recurrence of the tumor were recorded in the clinical assessments in the eCRF and not as SAE.
  Death due to a progressive disease were recorded on a specific form in the eCRF but not as a SAE.
Arm/Group | recMage-A3 + AS15 ASCI | Placebo
All-Cause Mortality (participants affected / at risk) | 6/48 | 5/29
Serious Adverse Events (participants affected / at risk) | 13/48 | 5/29
Other Adverse Events (participants affected / at risk) | 30/48 | 10/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | recMage-A3 + AS15 ASCI (N=48) | Placebo (N=29)
MASSIVE PROGRESSION OF LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
TACHYCARDIA VENTRICULAR (Cardiac disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
URINARY INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2)
STENOSIS OF GASTROINTESTINAL STOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIOGRAPHIC EVIDENCE OF CENTRAL TUMOR RENAL PELVIS LEFT (Investigations) | 1 (1) | 0 (0)
LOW BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PULMONARY CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
RIGHT URETERAL STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
LEFT URETERAL STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
PULMONARY THROMBOEMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
LEFT FEMORAL ATERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0)
PHLEBOTHROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | recMage-A3 + AS15 ASCI (N=48) | Placebo (N=29)
Influenza like illness (General disorders) | 5 (25) | 3 (6)
Injection site erythema (General disorders) | 4 (22) | 0 (0)
Injection site induration (General disorders) | 3 (21) | 0 (0)
Injection site pain (General disorders) | 17 (54) | 0 (0)
Pyrexia (General disorders) | 14 (41) | 4 (5)
Urinary tract infection (Infections and infestations) | 10 (11) | 5 (6)

LIMITATIONS AND CAVEATS:
Trial's recruitment was prematurely stopped. The recMAGE-A3+ AS15 patients were given the opportunity to continue treatment whereas placebo patients needed to stop treatment. All clinical data collected in this study were analysed descriptively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI submits the proposed publication to Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor shall have the right to remove from the proposed publication any information that is considered confidential and/or proprietary. Sponsor shall have the right to request an additional delay to the proposed disclosure of no more than ninety (90) days so as to allow Sponsor to preserve its intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT01435356/Prot_SAP_000.pdf